CLINICAL TRIAL: NCT02336113
Title: Oslo Pharmacist Intervention Study - Effect on Readmissions
Acronym: OPERA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Hospital Pharmacy Enterprise, South Eastern Norway (Other); South-Eastern Norway Regional Health Authority (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Morten Mowe, Associate professor, senior consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014/704
Record Dates: First submitted 2014-06-26; First posted 2015-01-12 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Acute Admitted Multimorbid Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Standard care during hospital stay, without pharmacist involved
- Pharmacist intervention (Experimental): A pharmacist is included in the multidisciplinary treatment team during the hospital stay
  Interventions: Behavioral: multidisciplinary treatment

INTERVENTIONS:
Behavioral: multidisciplinary treatment — The pharmacist will conduct medication reconciliation at admission, perform medication reviews during the hospital stay and provide drug information (written and oral) to the patient before discharge, as well as written drug information to the next level of care
  Arms: Pharmacist intervention

SUMMARY:
Earlier studies have shown that pharmacists detect and solve drug related problems (DRPs) when they are a part of the multidisciplinary treatment-team at hospital wards. However, in the Norwegian health care system, there is a lack of studies on the effect of pharmacist intervention on clinically relevant outcomes. Hospital readmissions has both clinical and economical negative effects, and time outside the hospital until an eventual readmission is considered as a clinical relevant outcome measure. The investigators are conducting a randomized controlled trial at an internal medicine ward at Oslo University Hospital. 400 acute admitted patients using minimum 4 regular drugs from minimum 2 drug groups will be enrolled in the study. Patients randomized to the Control group will receive standard care (without a pharmacist involved) and patients randomized to the Intervention group will receive a pharmacist in their treatment team during the hospital stay. The study hypothesis is that including a pharmacist in the multidisciplinary treatment team at a hospital ward, will improve the patients drug treatment, hence lead to an increased time outside the hospital until an eventual readmission.

The inclusion of patients was completed March 17th 2016 With 399 patients randomised. The last day of follow-up on readmission and mortality was December 31, 2017. The Application process for outcome data to the Norwegian Patient Registry and the Norwegian Cause of Death Registry started in June 2017 and lasted until May 2018. Huge workload at the Registers entails a very long processing time for outcome data. On May 25, 2018 the statistical analysis plan was finalized and signed, hereunder the analysis population defined and the endpoint analyses detailed. Outcome datafiles from patient registries was prepared for analysis May 29 to June 6, 2018. Blinded outcome analyses was conducted June 8, 2018.

_______________________________

The investigators have obtained approval for a protocol amendment to use the data from the study in further analyses togheter with data from 100 new patients admitted to the internal medicine ward. The hypothesis is that a set of patient characteristics can identify patients who are at high risk of drug-related readmissions and who would benefit most from the pharmaceutical intervention.The investigators aim to identify these patients by building a statistical model based on significant variables from the 399 patients collected in the randomised controlled trial. The statistical model will be validated using data from 100 new patients admitted to the internal medicine ward.

The inclusion of patients to this New sample was finalised July 6th 2018 (primary completion). Data on hospital readmissions and death will be collected from the Norwegian Patient Registry and the Norwegian Cause of Death Registry in June 2020.

ELIGIBILITY:
Inclusion Criteria:

* acute admitted patients using minimum 4 regular drugs from minimum 2 drug groups at admittance
* Norwegian personal identification number

Exclusion Criteria:

* terminally ill
* not able no communicate in Norwegian or English and an interpreter is not available
* patients isolated due to severe infections
* readmitted patients earlier included are not re-included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-07-06 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Days outside hospital until an eventual first readmission | 12 months after hospital discharge
  Calculated as the difference between the Control- and intervention group in the intention-to-treat population with data from The Norwegian Patient Register

CONTACTS AND LOCATIONS:
Overall Officials: Morten Mowe, Associate professor, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Lea M, Mowe M, Molden E, Kvernrod K, Skovlund E, Mathiesen L. Effect of medicines management versus standard care on readmissions in multimorbid patients: a randomised controlled trial. BMJ Open. 2020 Dec 29;10(12):e041558. doi: 10.1136/bmjopen-2020-041558. PMID 33376173